CLINICAL TRIAL: NCT00482677
Title: A Randomized Phase III Study of Temozolomide and Short-Course Radiation Versus Short-Course Radiation Alone In The Treatment of Newly Diagnosed Glioblastoma Multiforme in Elderly Patients
Brief Title: Radiation Therapy With or Without Temozolomide in Treating Older Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE6; CAN-NCIC-CE6 (Registry Identifier: NCI US - Physician Data Query); EORTC-26062-22061 (Other: EORTC); TROG 08.02 (Other: Trans-Tasman Radiation Oncology Group); SPRI-CAN-NCIC-CE.6; CDR0000547163 (Other: PDQ); NCT00493207 (obsolete NCT alias)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2020-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Temozolomide; DNA Methylation; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temozolomide (Active Comparator): Temozolomide and short course radiation
  Interventions: Drug: temozolomide; Genetic: DNA methylation analysis; Procedure: quality-of-life assessment
- Radiation (Active Comparator): Short course radiation alone
  Interventions: Genetic: DNA methylation analysis; Procedure: quality-of-life assessment; Radiation: Radiation

INTERVENTIONS:
Drug: temozolomide — Temozolomide (concurrent with radiation) 75 mg/m2 PO 3 weeks once a day, daily, from the first day to the last day of radiotherapy, but for no longer than 28 days, and then adjuvantly for up to 12 cycles (150 mg/m2 for the first 5 days of each cycle). Adjuvant TMZ may be escalated to 200mg/m2 in C2 onward if appropriate.
  Arms: Temozolomide
Genetic: DNA methylation analysis — A stratified log-rank test, adjusting for the stratification factors (except centre) plus MGMT promoter methylation status, will be used as the primary method to compare the overall survival between the two arms
Procedure: quality-of-life assessment — prior to randomization until end of study
Radiation: Radiation — Short course radiotherapy
  Arms: Radiation

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with temozolomide may kill more tumor cells. It is not yet known whether radiation therapy and temozolomide are more effective than radiation therapy alone in treating glioblastoma multiforme.

PURPOSE: This randomized phase III trial is studying radiation therapy and temozolomide to see how well they work compared with radiation therapy alone in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival rates in older patients with newly diagnosed glioblastoma multiforme treated with short-course radiotherapy with or without temozolomide.

Secondary

* Compare progression-free survival of patients treated with these regimens.
* Compare the nature, severity, and frequency of adverse events in patients treated with these regimens.
* Compare the quality of life of patient treated with these regimens.
* Determine the methylation status of the O6-methylguanine-DNA methyltransferase promoter.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to center, age (65-70 years vs 71-75 years vs ≥ 76 years), ECOG performance status (0-1 vs 2), and extent of resection at surgery (biopsy only vs complete or incomplete resection). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy once daily on days 1-5, 8-12, and 15-19 in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo radiotherapy as in arm I and receive oral temozolomide once daily on days 1-25.

Beginning 4 weeks after completion of radiotherapy and temozolomide, patients receive adjuvant oral temozolomide once daily on days 1-5. Treatment with temozolomide alone repeats every 28 days for up to 12 months in the absence of disease progression or unacceptable toxicity.

Patients complete quality of life questionnaires at baseline and periodically during study treatment.

Tissue samples are collected at baseline and analyzed for methylation status of the O6-methylguanine-DNA methyltransferase promoter.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically confirmed glioblastoma multiforme

  * Grade IV disease by WHO classification
  * Newly diagnosed disease
* Initial diagnostic surgery or biopsy performed within the past 4 weeks
* Not a candidate for standard radiotherapy (60Gy/30 fractions over 6 weeks) in combination with temozolomide

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* ALT and AST < 2.5 times ULN
* No known hypersensitivity to temozolomide or compounds with similar chemical composition to temozolomide
* No history of other malignancies except adequately treated nonmelanoma skin cancer, curatively treated in situ cancer of the cervix, or other curatively treated solid tumors with no evidence of disease for at least 5 years
* No serious active infection (e.g., wound infection requiring parenteral antibiotics) or other serious underlying medical conditions that would preclude study treatment
* No other condition (e.g., psychological or geographical) that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior radiotherapy
* No prior or concurrent investigational therapy
* No concurrent surgical procedures for tumor debulking
* No concurrent stereotactic boost radiotherapy
* No other concurrent chemotherapy, immunotherapy, or biological therapy
* No concurrent epoetin alfa
* Concurrent corticosteroids allowed provided the patient has been on a stable or decreasing dose for at least 14 days

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 562 (Actual)
Dates: Start 2007-11-14 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Normand Laperriere, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada; James R. Perry, MD, FRCPC, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Alba A. Brandes, MD, Study Chair — Ospedale Bellaria; Johan Menten, MD, PhD, Study Chair — University Hospital, Gasthuisberg
Locations (22):
- Canada (16):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec
- Germany (4):
  - Klinikum Der J.W. Goethe Universitaet, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Tuebingen, Tübingen
- Hiroshima University Hospital, Hiroshima, Japan
- Maastro - Maastricht Radiation Oncology, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perry JR, Laperriere N, O'Callaghan CJ, Brandes AA, Menten J, Phillips C, Fay M, Nishikawa R, Cairncross JG, Roa W, Osoba D, Rossiter JP, Sahgal A, Hirte H, Laigle-Donadey F, Franceschi E, Chinot O, Golfinopoulos V, Fariselli L, Wick A, Feuvret L, Back M, Tills M, Winch C, Baumert BG, Wick W, Ding K, Mason WP; Trial Investigators. Short-Course Radiation plus Temozolomide in Elderly Patients with Glioblastoma. N Engl J Med. 2017 Mar 16;376(11):1027-1037. doi: 10.1056/NEJMoa1611977. PMID 28296618
- [Derived] Climans SA, Brandes AA, Cairncross JG, Ding K, Fay M, Laperriere N, Menten J, Nishikawa R, O'Callaghan CJ, Perry JR, Phillips C, Roa W, Wick W, Winch C, Mason WP. Temozolomide and seizure outcomes in a randomized clinical trial of elderly glioblastoma patients. J Neurooncol. 2020 Aug;149(1):65-71. doi: 10.1007/s11060-020-03573-x. Epub 2020 Jul 6. PMID 32632894
- [Derived] Fiorentino A, De Bonis P, Chiesa S, Balducci M, Fusco V. Elderly patients with glioblastoma: the treatment challenge. Expert Rev Neurother. 2013 Oct;13(10):1099-105. doi: 10.1586/14737175.2013.840419. PMID 24117272

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide | Radiation
Started | 281 | 281
Completed | 281 | 281
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temozolomide | Radiation | Total
Number analyzed (Participants) | 281 | 281 | 562
Age, Continuous [Median (Full Range); unit: years] | 73 [65 to 90] | 73 [65 to 88] | 73 [65 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 109 | 219
  Male | 171 | 172 | 343
Region of Enrollment [Number; unit: participants]
  Canada | 101 | 98 | 199
  Netherlands | 48 | 49 | 97
  Japan | 8 | 9 | 17
  Germany | 124 | 125 | 249
ECOG Performance Status [Count of Participants; unit: Participants] — "The ECOG Scale of Performance Status ranges between 0 (Fully active, able to carry on all pre-disease performance without restriction) and 5 (Dead).
  Participants
    0, 1 | 215 | 217 | 432
    2 | 66 | 64 | 130
Resection [Count of Participants; unit: Participants]
  Biopsy only | 84 | 82 | 166
  Complete/incomplete resection | 197 | 199 | 396
Mini Mental Status Examination [Median (Full Range); unit: participants] | 27 [5 to 30] | 27 [7 to 30] | 27 [5 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from date of randomization to the date of death of any causes, or censored at last known alive date.
Time Frame: 7 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Temozolomide | Radiation
Number analyzed (Participants) | 281 | 281
Months | 9.33 [8.31 to 10.25] | 7.62 [6.97 to 8.38]

2. Secondary Outcome: Progression-free Survival
Description: Time from date of randomization to the date of disease progression or death whichever came first, or censored at last disease assessment date.
Time Frame: 7 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Temozolomide | Radiation
Number analyzed (Participants) | 281 | 281
Months | 5.29 [4.60 to 6.21] | 3.94 [3.52 to 4.34]

3. Secondary Outcome: Adverse Events
Description: Evaluated according to CTCAE V3.0
Time Frame: 7 years
Reporting Status: Not Posted

4. Secondary Outcome: Methylation Status of the O6-methylguanine-DNA Methyltransferase Promoter
Description: Overall survival for patients by Methylation status of the O6-methylguanine-DNA methyltransferase promoter
Time Frame: 7 years
Population: Patients with MGMT promoter methylated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Temozolomide | Radiation
Number analyzed (Participants) | 88 | 77
Months | 13.47 [10.25 to 15.31] | 7.69 [5.82 to 10.68]

ADVERSE EVENTS:
Arm/Group | Temozolomide | Radiation
Serious Adverse Events (participants affected / at risk) | 158/271 | 135/271
Other Adverse Events (participants affected / at risk) | 260/271 | 256/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide (N=271) | Radiation (N=271)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1 | 2
Cardiopulmonary arrest (Cardiac disorders) | 2 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Pain Cardiac/heart (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia Atrial fibrillation (Cardiac disorders) | 2 | 1
Ventricular arrhythmia Ventricular tachycardia (Cardiac disorders) | 1 | 0
Blurred vision (Eye disorders) | 2 | 1
Glaucoma (Eye disorders) | 1 | 0
Neuropathy: cranial CN II (Eye disorders) | 2 | 3
Pain Eye (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 7 | 5
Hemorrhage, GI Lower GI NOS (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI Rectum (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Incontinence, anal (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Pain Abdomen NOS (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Perforation, GI Colon (Gastrointestinal disorders) | 2 | 1
Perforation, GI Esophagus (Gastrointestinal disorders) | 1 | 0
Ulcer, GI Stomach (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2
Constitutional Symptoms - Other (General disorders) | 1 | 1
Death Death NOS (General disorders) | 7 | 7
Death Disease progression NOS (General disorders) | 1 | 3
Edema: head and neck (General disorders) | 1 | 3
Edema: limb (General disorders) | 1 | 1
Fatigue (General disorders) | 17 | 16
Fever (General disorders) | 5 | 3
Gait/walking (General disorders) | 1 | 1
Pain Pain NOS (General disorders) | 0 | 1
Syndromes - Other (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Infection (documented clinically) Colon (Infections and infestations) | 1 | 0
Infection (documented clinically) Lung (Infections and infestations) | 2 | 4
Infection (documented clinically) Muscle (Infections and infestations) | 1 | 0
Infection (documented clinically) Peritoneal cavity (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 2 | 2
Infection with normal ANC Abdomen NOS (Infections and infestations) | 1 | 0
Infection with normal ANC Bladder (Infections and infestations) | 0 | 1
Infection with normal ANC Blood (Infections and infestations) | 4 | 0
Infection with normal ANC Brain (Infections and infestations) | 1 | 0
Infection with normal ANC Colon (Infections and infestations) | 1 | 0
Infection with normal ANC Lung (Infections and infestations) | 6 | 2
Infection with normal ANC Peritoneal cavity (Infections and infestations) | 1 | 0
Infection with normal ANC Skin (Infections and infestations) | 0 | 1
Infection with normal ANC Soft tissue NOS (Infections and infestations) | 0 | 1
Infection with normal ANC Upper airway NOS (Infections and infestations) | 0 | 1
Infection with normal ANC Urinary tract NOS (Infections and infestations) | 1 | 1
Infection with normal ANC Wound (Infections and infestations) | 1 | 1
Infection with unknown ANC Blood (Infections and infestations) | 1 | 0
Infection with unknown ANC Bronchus (Infections and infestations) | 1 | 0
Infection with unknown ANC Lung (Infections and infestations) | 1 | 3
Infection with unknown ANC Skin (Infections and infestations) | 0 | 1
Infection with unknown ANC Urinary tract NOS (Infections and infestations) | 1 | 0
Dermatitis Radiation (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 6 | 7
Thrombosis/embolism (vascular access) (Injury, poisoning and procedural complications) | 3 | 2
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 | 0
ADH (Investigations) | 0 | 1
GGT (Investigations) | 1 | 0
Platelets (Investigations) | 4 | 2
Weight loss (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Diabetes (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Joint-function (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness Extremity-lower (Musculoskeletal and connective tissue disorders) | 8 | 2
Muscle weakness Extremity-upper (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness Left-sided (Musculoskeletal and connective tissue disorders) | 3 | 4
Muscle weakness Right-sided (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle weakness Whole body/generalized (Musculoskeletal and connective tissue disorders) | 5 | 5
Pain Back (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain Bone (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Arachnoiditis (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 6 | 6
CNS hemorrhage (Nervous system disorders) | 2 | 2
CNS ischemia (Nervous system disorders) | 5 | 2
CNS necrosis (Nervous system disorders) | 0 | 1
CSF leak (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 16 | 11
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 3 | 0
Involuntary movement (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 3
Neurology - Other (Nervous system disorders) | 2 | 3
Neuropathy-motor (Nervous system disorders) | 29 | 22
Neuropathy-sensory (Nervous system disorders) | 1 | 3
Neuropathy: cranial CN III (Nervous system disorders) | 1 | 0
Neuropathy: cranial CN VII (Nervous system disorders) | 1 | 0
Neuropathy: cranial CN VIII (Nervous system disorders) | 0 | 1
Pain Head/headache (Nervous system disorders) | 5 | 7
Pyramidal tract dysfunction (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 27 | 20
Somnolence (Nervous system disorders) | 11 | 20
Speech impairment (Nervous system disorders) | 16 | 21
Syncope (Nervous system disorders) | 1 | 3
Confusion (Psychiatric disorders) | 17 | 23
Mood alteration Agitation (Psychiatric disorders) | 7 | 3
Mood alteration Anxiety (Psychiatric disorders) | 1 | 1
Mood alteration Depression (Psychiatric disorders) | 4 | 1
Personality (Psychiatric disorders) | 0 | 2
Psychosis (Psychiatric disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 0 | 1
Hemorrhage, GU Kidney (Renal and urinary disorders) | 1 | 0
Incontinence, urinary (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Hemorrhage, GU Prostate (Reproductive system and breast disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Hemorrhage pulmonary Nose (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatology - Other (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Phlebitis (Vascular disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 25 | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide (N=271) | Radiation (N=271)
Hearing (without monitoring program) (Ear and labyrinth disorders) | 15 | 14
Blurred vision (Eye disorders) | 15 | 21
Constipation (Gastrointestinal disorders) | 74 | 29
Diarrhea (Gastrointestinal disorders) | 19 | 5
Dysphagia (Gastrointestinal disorders) | 20 | 18
Nausea (Gastrointestinal disorders) | 77 | 42
Vomiting (Gastrointestinal disorders) | 38 | 15
Edema: limb (General disorders) | 50 | 35
Fatigue (General disorders) | 158 | 147
Gait/walking (General disorders) | 22 | 19
Dermatitis Radiation (Injury, poisoning and procedural complications) | 22 | 22
Anorexia (Metabolism and nutrition disorders) | 41 | 38
Muscle weakness Extremity-lower (Musculoskeletal and connective tissue disorders) | 42 | 34
Muscle weakness Whole body/generalized (Musculoskeletal and connective tissue disorders) | 17 | 18
Pain Muscle (Musculoskeletal and connective tissue disorders) | 16 | 8
Ataxia (Nervous system disorders) | 30 | 29
Cognitive disturbance (Nervous system disorders) | 55 | 46
Dizziness (Nervous system disorders) | 43 | 25
Memory impairment (Nervous system disorders) | 66 | 64
Neurology - Other (Nervous system disorders) | 19 | 16
Neuropathy-motor (Nervous system disorders) | 77 | 65
Neuropathy-sensory (Nervous system disorders) | 24 | 15
Pain Head/headache (Nervous system disorders) | 64 | 78
Seizure (Nervous system disorders) | 73 | 57
Somnolence (Nervous system disorders) | 24 | 39
Speech impairment (Nervous system disorders) | 68 | 77
Tremor (Nervous system disorders) | 18 | 16
Confusion (Psychiatric disorders) | 66 | 65
Insomnia (Psychiatric disorders) | 31 | 31
Mood alteration Agitation (Psychiatric disorders) | 26 | 16
Mood alteration Anxiety (Psychiatric disorders) | 19 | 12
Mood alteration Depression (Psychiatric disorders) | 37 | 20
Incontinence, urinary (Renal and urinary disorders) | 22 | 17
Urinary frequency (Renal and urinary disorders) | 19 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 27
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30 | 25
Alopecia (Skin and subcutaneous tissue disorders) | 69 | 77
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 8
Rash (Skin and subcutaneous tissue disorders) | 29 | 19
Thrombosis/thrombus/embolism (Vascular disorders) | 34 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No